CLINICAL TRIAL: NCT05839665
Title: Evaluation of Different Methods for Preoxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malin Jonsson Fagerlund (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Malin Jonsson Fagerlund, Associate Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PreFlow
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia
Keywords: Preoxygenation; Oxygenation; High-flow nasal oxygen; Low-flow nasal oxygen

STUDY DESIGN:
Intervention Model Description: All volunteers will start with pre-oxygenation using a traditional facemask (vital breathing for four minutes vital and eight vital capacity breaths). They will thereafter be randomised to continue with either pre-oxygenation using a standard nasal cannula or humidified high-flow nasal oxygen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Humidified high-flow oxygen (Active Comparator): Humidified high-flow nasal oxygen delivered via the Optiflow device. Repeated series with 100% oxygen with flows varying between 30 to 50 l/min. Volunteers will also be pre-oxygenated with both opened and closed mouth.
  Interventions: Device: Humidified high-flow nasal oxygen
- Standard nasal cannula (Experimental): Standard nasal cannula connected to an oxygen rotameter Repeated series with 100% oxygen with flows varying between 15 to 50 l/min. Volunteers will also be pre-oxygenated with both opened and closed mouth.
  Interventions: Device: Standard nasal cannula
- Facemask (Active Comparator): Tight-fitting facemask. Two series will be done where pre-oxygenation will be performed with four minutes of tidal volume breathing and eight vital capacity breaths.
  This arm is not randomised. All study subjects will start with facemask pre-oxygenation and are thereafter randomised to standard nasal cannula or humidified high-flow nasal cannula.
  Interventions: Device: Facemask

INTERVENTIONS:
Device: Humidified high-flow nasal oxygen — Humidified high-flow oxygen delivered via the Optiflow device
  Arms: Humidified high-flow oxygen
Device: Standard nasal cannula — Oxygen delivered with high flows via a standard nasal cannula
  Arms: Standard nasal cannula
Device: Facemask — Oxygen delivered with facemask
  Arms: Facemask

SUMMARY:
The goal of this randomised cross-over study is to compare pre-oxygenation using a standard nasal cannula to pre-oxygenation using humidified high-flow nasal oxygen and a tight-fitting facemask in adult volunteers with a BMI below 30 not suffering from pulmonary or cardiac comorbidity.

The main question it aims to answer is:

- Are there any differences in the effectiveness of pre-oxygenation using a standard nasal cannula compared to using a traditional facemask and pre-oxygenation using humidified high-flow nasal oxygen?

Participants will be pre-oxygenated with 100% oxygen during four minutes intervals. All participants will be pre-oxygenated with various flow rates using a standard nasal cannula, a facemask and humidified high-flow nasal oxygen. End-tidal oxygen concentrations will be measured continuously in order to evaluate the effectiveness of pre-oxygenation.

Each volunteer will be pre-oxygenated repeatedly, with different flow rates, with all three methods of pre-oxygenation and act as its own control.

During facemask pre-oxygenation volunteers will be pre-oxygenated using both tidal volume breathing for four minutes and with eight vital capacity breaths. During pre-oxygenation using the standard nasal cannula flow rates will vary between 15 and 50 l/min. Pre-oxygenation using humidified high-flow nasal oxygen will be performed with flow rates varying between 30 and 50 l/min. Series will be conducted with volunteers breathing with both opened and closed mouth as well as with four minutes of tidal volume breathing and eight vital capacity breaths.

All volunteers will start with facemask pre-oxygenation. They will thereafter be randomised to pre-oxygenation with either a standard nasal cannula or humidified high-flow nasal oxygen. Lastly, they will be pre-oxygenated with the remaining method according to the randomisation.

DETAILED DESCRIPTION:
Pre-oxygenation before anaesthesia induction is mostly performed using a tight-fitting facemask. Recently, studies have shown that pre-oxygenation using humidified high-flow nasal oxygen is equally effective as pre-oxygenation using a standard tight-fitting facemask. Pre-oxygenation using humidified high-flow nasal oxygen has several potential advantages including improved patient comfort and the possibility of a seamless transition from pre-oxygenation to apnoeic oxygenation. Unfortunately, this technique requires an additional machine which can be expensive and also difficult to use in settings outside a hospital.

In this study, pre-oxygenation using a standard nasal cannula delivering a high flow of oxygen will be compared with standard facemask pre-oxygenation and pre-oxygenation using humidified high-flow nasal oxygen in adult volunteers with a BMI below 30 not suffering from pulmonary or cardiac comorbidity.

The main question it aims to answer is:

- Are there any differences in the effectiveness of pre-oxygenation using a standard nasal cannula compared to using a traditional facemask and pre-oxygenation using humidified high-flow nasal oxygen?

Participants will be pre-oxygenated with 100% oxygen during four minutes intervals. All participants will be pre-oxygenated with various flow rates using a standard nasal cannula, a facemask and humidified high-flow nasal oxygen. End-tidal oxygen concentrations will be measured continuously in order to evaluate the effectiveness of pre-oxygenation.

Each volunteer will be pre-oxygenated repeatedly, with different flow rates, with all three methods of pre-oxygenation and act as its own control.

During facemask pre-oxygenation volunteers will be pre-oxygenated using both tidal volume breathing for four minutes and with eight vital capacity breaths. During pre-oxygenation using the standard nasal cannula flow rates will vary between 15 and 50 l/min. Pre-oxygenation using humidified high-flow nasal oxygen will be performed with flow rates varying between 30 and 50 l/min. Series will be conducted with volunteers breathing with both opened and closed mouth as well as with four minutes of tidal volume breathing and eight vital capacity breaths.

All volunteers will start with facemask pre-oxygenation. They will thereafter be randomised to pre-oxygenation with either a standard nasal cannula or humidified high-flow nasal oxygen. Lastly, they will be pre-oxygenated with the remaining method according to the randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign informed consent
* Age 25-65 years
* Body mass index <30

Exclusion Criteria:

* Heart disease
* Respiratory disease
* Pregnancy
* Smoker

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the effectiveness of pre-oxygenation | After 3 minutes of preoxygenation
  Compare end-tidal oxygen levels after three minutes of pre-oxygenation using a standard facemask, high-flow nasal oxygen and a standard nasal cannula.

SECONDARY OUTCOMES:
Duration of pre-oxygenation until end-tidal oxygen levels above 80% | After 3 minutes of preoxygenation
  Evaluation of end-tidal oxygen levels will be done each minute during all series of pre-oxygenation in order to investigate the time taken until reaching end-tidal levels above 80%. A comparison between the time taken to achieve end-tidal levels above 80% will be done between the different methods of pre-oxygenation as well as the different flow rates.
Duration of pre-oxygenation until end-tidal oxygen levels above 85% | After 3 minutes of preoxygenation
  Evaluation of end-tidal oxygen levels will be done each minute during all series of pre-oxygenation in order to investigate the time taken until reaching end-tidal levels above 85%. A comparison between the time taken to achieve end-tidal levels above 80% will be done between the different methods of pre-oxygenation as well as the different flow rates.
Continuous comparison of end-tidal oxygen levels | After 3 minutes of preoxygenation
  Evaluation of end-tidal oxygen levels will be done after one, two, three and four minutes of pre-oxygenation. Comparison between the different methods and flow rates of pre-oxygenation will be done in order to evaluate which method and flow rate generates adequate end-tidal oxygen levels most quickly.
Pre-oxygenation with open and closed mouth | After 3 minutes of preoxygenation
  All volunteers will be pre-oxygenated with both open and closed mouths in order to evaluate if there are any differences in end-tidal oxygen levels when breathing with open or closed mouth.
Vital capacity breathing vs tidal volume breathing | After 3 minutes of preoxygenation
  End-tidal oxygen levels during pre-oxygenation will be evaluated and compared between tidal volume breathing for three minutes and eight vital capacity breaths.
Differences in end-tidal oxygen levels after pre-oxygenation due to age, body mass index or sex. | After 3 minutes of preoxygenation
  Subgroup analysis will be performed in order to investigate any differences in the effect of pre-oxygenation depending on volunteer age, body mass index or sex.
Discomfort | After 3 minutes of preoxygenation
  Level of discomfort, on a scale between one and ten, where ten is the worst discomfort and 0 is the best comfort) will be compared between the three different methods of pre-oxygenation and the different flow rates.

OTHER OUTCOMES:
Safety outcome | After 3 minutes of preoxygenation
  Do more volunteers report problem with headache or nosebleed during pre-oxygenation with the standard nasal cannula compared to pre-oxygenation with facemask or humidified high-flow nasal oxygen?

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, Principal Investigator — Karolinska University Hospital and Karolinska Institutet
Locations (2):
- Sweden (2):
  - Perioperative Medicine and Intensive Care Medicine, Stockholm
  - Karolinska University Hospital, Solna, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sjoblom A, Hedberg M, Forsberg IM, Hoffman F, Jonsson Fagerlund M. Comparison of preoxygenation using a tight facemask, humidified high-flow nasal oxygen and a standard nasal cannula - a volunteer, randomised, crossover study. Eur J Anaesthesiol. 2024 Jun 1;41(6):430-437. doi: 10.1097/EJA.0000000000001989. Epub 2024 Apr 16. PMID 38630525